CLINICAL TRIAL: NCT00912509
Title: A Prospective Randomized Double-masked Evaluation of Treatment Duration of the UVX System for Treating Infectious Keratitis
Brief Title: Cross Linking for Treatment of Corneal Infection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient efficacy
Sponsor: Price Vision Group (Industry)
Collaborators: Cornea Research Foundation of America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-0143
Record Dates: First submitted 2009-05-30; First posted 2009-06-03 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-10

CONDITIONS: Infectious Keratitis
Keywords: infectious keratitis; cross linking; corneal ulcer; corneal infection; collagen cross linking
MeSH Terms: conditions — Corneal Ulcer | interventions — Riboflavin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 30 minute light duration (Active Comparator): 30 minute treatment with UVX light
  Interventions: Drug: riboflavin; Device: UVX Light
- 45 minute light duration (Active Comparator): 45 minute treatment with UVX light
  Interventions: Device: UVX Light

INTERVENTIONS:
Drug: riboflavin — riboflavin 0.1% is applied every 2 minutes for 30 minutes
  Arms: 30 minute light duration
Device: UVX Light — UVX 365 nm wavelength light source is applied with continued application of riboflavin 0.1%

SUMMARY:
This study is comparing 45 minute and 30 minute treatment durations with the UVX corneal cross linking system to treat corneal infections.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of infectious keratitis

Exclusion Criteria:

* corneal ulcer that has perforated
* corneal ulcer that has produced a descemetocele
* women who are pregnant or breastfeeding
* patients who are immunocompromised or unwilling or unable to comply with a medication regimen

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis W Price, MD, Principal Investigator — Price Vision Group
Locations (1):
- Price Vision Group, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Iseli HP, Thiel MA, Hafezi F, Kampmeier J, Seiler T. Ultraviolet A/riboflavin corneal cross-linking for infectious keratitis associated with corneal melts. Cornea. 2008 Jun;27(5):590-4. doi: 10.1097/ICO.0b013e318169d698. PMID 18520510
- [Result] Price MO, Tenkman LR, Schrier A, Fairchild KM, Trokel SL, Price FW Jr. Photoactivated riboflavin treatment of infectious keratitis using collagen cross-linking technology. J Refract Surg. 2012 Oct;28(10):706-13. doi: 10.3928/1081597X-20120921-06. PMID 23062001
- [Derived] Davis SA, Bovelle R, Han G, Kwagyan J. Corneal collagen cross-linking for bacterial infectious keratitis. Cochrane Database Syst Rev. 2020 Jun 17;6(6):CD013001. doi: 10.1002/14651858.CD013001.pub2. PMID 32557558
- See also: Price Vision Group website — http://www.pricevisiongroup.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 30 Minute Light Duration | 45 Minute Light Duration
Started | 20 | 10
Completed | 15 | 7
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Lack of Efficacy | 4 | 3

BASELINE CHARACTERISTICS:
Population: This is the number of participants who were culture-positive
Groups:
- 45 Minute Light Duration: 45 minute treatment with UVX light
  riboflavin: riboflavin 0.1% is applied every 2 minutes for 30 minutes
  UVX Light: UVX 365 nm wavelength light source is applied with continued application of riboflavin 0.1%
- Total: Total of all reporting groups
Arm/Group | 30 Minute Light Duration | 45 Minute Light Duration | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 13 | 4 | 17
  >=65 years | 6 | 6 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 6 | 20
  Male | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Time to Re-epithelialization
Time Frame: Day 1, day 2, day 3, day 4, day 5, day 6, day 7, week 2, and subsequent weekly assessments until re-epithelialization is complete
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | 30 Minute Light Duration | 45 Minute Light Duration
Number analyzed (Participants) | 15 | 7
Days | 14 [6 to 28] | 11 [6 to 29]

2. Secondary Outcome: Time to Resolution of Stromal Infiltration
Time Frame: day 1, day 2, day 3, day 4, day 5, day 6, day 7, week 2, and subsequent weekly assessments until infiltrate is completely resolved
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | 30 Minute Light Duration | 45 Minute Light Duration
Number analyzed (Participants) | 15 | 7
days | 21 [8 to 33] | 10 [7 to 11]

ADVERSE EVENTS:
Arm/Group | 30 Minute Light Duration | 45 Minute Light Duration
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 5/20 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 30 Minute Light Duration (N=20) | 45 Minute Light Duration (N=10)
Cornea transplant (Eye disorders) | 4 (4) | 2 (2)
Intracorneal injection of voriconazole (Eye disorders) | 1 (1) | 1 (1)
Dendritic lesions characteristic of prior herpes simplex (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No